CLINICAL TRIAL: NCT06690749
Title: Effect of Negative Pressure Therapy on Skin Blood Flow Responses in the Scar
Brief Title: Using Skin Blood Flow to Measure the Effect of Different Doses of Negative Pressure Therapy
Acronym: Negative press
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRREC-111-017; NSTC 112-2221-E-468-004 (Other: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2024-11-05; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2022-05

CONDITIONS: Hypertrophic Scars
Keywords: Scar; Laser Doppler; Tensile stresses; Capillaries; Cupping
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Intervention Model Description: The study design and setting sample were drawn from patients randomly assigned to one of three parallel groups, initially in a 1:1:1 ratio to invite the subject to receive either NPT dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Negative pressure therapy dosage (Experimental): A negative pressure value gap of 20mmHg was used between the each groups.
  Interventions: Device: Negative pressure therapy, NPT

INTERVENTIONS:
Device: Negative pressure therapy, NPT — We designed the experiment based on current clinical cases involving negative pressure therapy (NPT) for wounds and related animal studies. In this study, we applied three levels of negative pressure: -105 mmHg, -125 mmHg, and -145 mmHg, each for 10 minutes.
  The -125 mmHg dosage was chosen based on findings from a previous study. Similar studies that utilized increments and decrements of 20 mmHg informed our research.
  Moreover, to prevent any damage to new capillaries, we established a base dosage of -125 mmHg and refrained from using negative pressure levels exceeding -150 mmHg.
  Other Names: -105 mmHg NPT; -125 mmHg NPT; -145 mmHg NPT

SUMMARY:
Introduction. Skin blood flow (SBF) is crucial for transporting nutrients during healing to treat scarring. Negative pressure therapy (NPT) is a promising option to enhance SBF. However, it is unclear what dosage of NPT is most effective in treating scars.

This study compared NPT dosages of -105 mmHg, -125 mmHg, and -145 mmHg to assess the impact of NPT treatment on SBF in scar tissue and the correlation of NPT. If participants experience any symptoms of discomfort, NPT can be discontinued immediately.

36 scarred subjects were recruited to assess the efficacy of various NPT interventions. SBF applications are defined as perfusion levels instantly affecting NPT, and termination is defined as SBF after NPT.

The study runs from May 11, 2022, to May 11, 2023, at Asia University Hospital.

This study was funded by the National Science and Technology Council, Taiwan (NSTC 112-2221-E-468-004)

The main contact was Chi-Wen Lung, the person in charge of a college or university department of Product Design, Asia University, Taichung 413305, Taiwan.Email address: cwlung@asia.edu.tw

DETAILED DESCRIPTION:
Introduction. Skin blood flow (SBF) is crucial for transporting nutrients during healing to treat scarring. Negative pressure therapy (NPT) is a promising option to enhance SBF.

This study's hypothesis was that NPT can enhance SBF in scar tissue and that the specific NPT dose affects this effect. The purpose of this study was to confirm the different dosages of NPT applied to scar tissue by comparing the blood flow before and after the effects of different NPT dosages. This will also contribute to the emerging field of scar treatment and provide evidence-based recommendations.

All recruited participants were approached to participate in a research study investigating the effects of NPT in a double-blind, parallel-group study on scar healing. This study used three negative pressure changes at -105, -125 mmHg, and -145 mmHg at 10 min. The suction method created a negative pressure in the cup using an electronic negative-pressure device (Medi Pump TC-2000V; Anest Iwata Sparmax Co., Ltd., Taipei, Taiwan). A cup with an inner diameter of 45 mm and outer diameter of 53 mm was used for cupping therapy. Each side of the cup rim had a width of 4 mm; therefore, no pain was caused by the cup rim.

Pearson product-moment correlation analysis was used to determine the correlations between the SBF-Baseline, SBF-Application, and SBF-Termination factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Wounds must have been present for at least 21 days.
* The participants were in the proliferation or remodeling phase.
* Within nine months of skin injury.

Exclusion Criteria:

* Incomplete wound healing.
* leakage of tissue fluid.
* Participants of the Edema.
* The other short-term treatment plans (pressure garments, radiotherapy, steroids, and cryotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Skin Blood Flow | Three minutes before to three minutes after negative pressure treatment
  The skin blood flow (SBF) before negative pressure therapy (NPT) recorded from 30 seconds to 1 minute was defined as the SBF-termination value.
  The 0-30 seconds SBF before NPT was the baseline SBF-Baseline. The records of the calculated NPT value from 10 minutes to 10.5 min are defined as application value.
  The record with 30 seconds to 1 minute after NPT is defined as the SBF-termination value. The evaluation standard is the 30-second average.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The raw data values of the skin blood flow study result in the Clinical Study Report (CSR) will be provided to the submitting journal when the relevant journal publishes.